CLINICAL TRIAL: NCT03385057
Title: Postoperative Ibuprofen Use and Risk of Bleeding in Pediatric Tonsillectomy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study design flaws; research design needed to be reconfigured
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Emory University (Other); University Hospitals Cleveland Medical Center (Other); Madigan Army Medical Center (U.S. Federal Agency); United States Naval Medical Center, Portsmouth (U.S. Federal Agency); Rady Children's Hospital, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-167H
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Tonsillectomy With or Without Adenoidectomy
MeSH Terms: interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibuprofen Arm (Active Comparator)
  Interventions: Drug: Ibuprofen
- Acetaminophen (Active Comparator)
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Ibuprofen — Grape-flavored ibuprofen 100mg/5mL (Leader®) will be dispensed. Ibuprofen will be dosed at 10mg/kg (max dose 600mg) QID (roughly Q6 hours, however we left dosing QID to allow for some flexibility in the dosing schedule to accommodate patient sleeping schedules). The pharmacy will manipulate the volume of each medication using Ora Blend suspension so that for each child, weight-based dosing of each medication will be equivalent in volume. The first dose of study medication will be dispensed 4 hours after the preoperative acetaminophen dose. Thereafter, medication will be dosed QID (or roughly 6 hours apart). Surgeons, nursing staff, and patients and their families will be blinded regarding the type of medication administered.
  Other Names: Motrin
  Arms: Ibuprofen Arm
Drug: Acetaminophen — Grape-flavored acetaminophen 160mg/5mL (Leader®) will be dispensed based upon the arm to which each participant has been randomized. Acetaminophen at 15mg/kg (max dose 650mg), dosing will be QID (roughly Q6 hours, however we left dosing QID to allow for some flexibility in the dosing schedule to accommodate patient sleeping schedules). The pharmacy will manipulate the volume of each medication using Ora Blend suspension so that for each child, weight-based dosing of each medication will be equivalent in volume. The first dose of study medication will be dispensed 4 hours after the preoperative acetaminophen dose. Thereafter, medication will be dosed QID (or roughly 6 hours apart). Surgeons, nursing staff, and patients and their families will be blinded regarding the type of medication administered.
  Other Names: Advil
  Arms: Acetaminophen

SUMMARY:
Pediatric tonsillectomy is one of the most common surgical procedures annually in the United States; risks include postoperative hemorrhage and poor pain control. Controversy exists regarding optimal pharmacologic pain management following surgery, as each drug's efficacy is balanced by its specific side effects. Ibuprofen is effective in controlling postoperative pain following tonsillectomy, but its mechanism of action results in decreased platelet function, which may increase postoperative bleeding events. This is a multicenter, randomized control non-inferiority trial designed to assess the relationship between short-course ibuprofen use and post-tonsillectomy bleeding when compared to acetaminophen.

DETAILED DESCRIPTION:
Pediatric tonsillectomy is one of the most common surgical procedures in the United States, with over 500,000 procedures performed annually.1,2 The most common indications for tonsillectomy with and without adenoidectomy are sleep-disordered breathing and recurrent tonsillitis, though significant demographic and regional variation exist.2 In recent years, particular attention has been paid to the deleterious sequelae of pediatric obstructive sleep apnea on children's behavior, cognition, and growth as well as its negative effects on long-term pulmonary and cardiovascular health.3-5 Tonsillectomy is generally considered a safe procedure, though potential exists for significant procedural morbidity. Potential risks associated with tonsillectomy include postoperative hemorrhage, airway risk, aspiration, burn injury, post-operative nausea and vomiting, and poor pain control.6,7 Postoperative hemorrhage is the most serious post-tonsillectomy complication and can be divided according to timing (primary occurring <24 hours from surgery, or secondary occurring >24 hours after surgery) and severity (level 1: any history of bleeding, level 2: bleeding requiring inpatient admission, level 3: bleeding requiring operative intervention). Following discharge, inadequate analgesia can result in secondary complications such as dehydration, nausea, bleeding, hospital readmission, and increased healthcare expenditures.8,9

Significant controversy exists as to the optimal pain management protocol following pediatric tonsillectomy.8,9 Many studies have examined both pharmacologic and non-pharmacologic modalities to improve pain control in this population. The most common medications prescribed after tonsillectomy include acetaminophen (paracetamol), non-steroidal anti-inflammatory drugs (NSAIDs) (e.g. ibuprofen), and narcotic pain medications, each with a unique mode of action and risk profile.8,10-12 Acetaminophen, which has both peripheral and central anti-nociceptive properties, is generally well-tolerated with low incidence of serious side effects, but may not provide adequate pain control when used at recommended pediatric dosages.13 Narcotic (opioid) pain medications act on the mu opioid receptor and effectively decrease sensory and affective components of pain.14 Unfortunately, opioid pain medications also result in dose-dependent respiratory depression; a significant contraindication in patients with sleep-disordered breathing.15,16 The FDA has released a warning cautioning against the use of codeine, an opioid, for postoperative analgesia following tonsillectomy.7 Furthermore, emerging data suggests that adolescent patients receiving prescription for narcotic pain medication may be at risk for long-term opioid dependence and addiction.17 NSAIDs provide analgesia through reversible COX-1 and COX-2 pathway inhibition which results in decreased prostaglandin-induced inflammation and edema.18 This mechanism of action also interferes with platelet aggregation, potentially impacting bleeding in the postoperative period. Ibuprofen, a derivative of propionic acid, is one of the most commonly prescribed NSAID medications, with a half-life of less than 12 hours.19,20 Pain control in patients receiving NSAIDs is equivalent, or superior to, those receiving acetaminophen alone or in combination with narcotic medication.21-23 In 2011, the American Academy of Pediatrics released its Clinical Practice Guidelines, which stated that ibuprofen can safely be used for postoperative analgesia following tonsillectomy24, a recommendation based on a 2005 Cochrane Review of NSAIDs and post-tonsillectomy bleeding. The most recent Cochrane review on this topic, published in 2012 and based on 15 randomized control trials (RCTs), concludes that there is insufficient evidence available to exclude an increased risk of bleeding with NSAID use following pediatric tonsillectomy.25 This is supported by data from a prospective, randomized control non-inferiority trial conducted at our own institution, in which participants received either ibuprofen or acetaminophen for 9 days following surgery. In this study, an increased rate of post-tonsillectomy bleeding requiring operative intervention could not be excluded because the non-inferiority threshold was crossed. The duration of safe NSAID use, if any, after tonsillectomy is unknown. A study definitively documenting safety and efficacy of short-course NSAID administration following tonsillectomy in children would affect our own standard of care as well as overall clinical practice guidelines.

This study serves as a follow-up clinical trial to a double-blind randomized control non-inferiority trial titled "Postoperative Ibuprofen and the Risk of Bleeding After Tonsillectomy with or without Adenoidectomy" conducted from 2012 to 2016 at Massachusetts Eye and Ear and collaborating institutions. In this study, participants were randomized to receive either ibuprofen (10 mg/kg every 6 hours) or acetaminophen (15 mg/kg every 6 hours) for 9 days following surgery. The non-inferiority margin was set at 3%. Increased type 3 bleeding (bleeding requiring operative intervention) could not be excluded because the non-inferiority threshold was crossed.

In this study, type 3 bleeding occurred in the ibuprofen group on an average postoperative day of 5.95. Additional analyses were conducted on study subjects who discontinued the study drugs prior to postoperative day 9 (the scheduled end point). A total of 50 patients discontinued study medication on or before postoperative day 3. Of these, 21 were randomized to the ibuprofen arm and 0/21 experienced postoperative bleeding events.

A recent systematic review by Tan et al examined commonly used medications following tonsillectomy and efficacy and risks associated with each drug.8 Acetaminophen is commonly used following tonsillectomy given its low side effect profile; however, analgesia is often inadequate at recommended dosages.26 Despite a 2013 FDA warning cautioning against opioid use following pediatric tonsillectomy due to increased risk of respiratory depression, these medications continue to be prescribed following surgery. The majority of tonsillectomies are now performed for sleep apnea and sleep disordered breathing; therefore, a large proportion of patients have increased risk of respiratory compromise and desaturations following surgery when opioid medications are administered.22 Furthermore, emerging data suggests that a significant fraction of adolescent patients receiving opioid pain medications postoperatively may subsequently develop addiction to these medications.17 NSAIDs are effective for post-tonsillectomy analgesia, but concerns remain regarding increased risk of postoperative hemorrhage with use of these medications despite current American Academy of Pediatrics recommendations advocate that ibuprofen may be safely utilized following tonsillectomy in children. Studies to date demonstrate conflicting or equivocal results with regard to increased bleeding risk following NSAID administration. Given previous data from this institution which cannot exclude increased incidence of type 3 bleeding following 9 days of ibuprofen exposure, MEE standard of practice is to recommend against extended duration of ibuprofen use in the postoplerative period. However, given concerns of inadequate analgesia with acetaminophen and respiratory depression and addictive potential with opioid medication, we feel that it is important to assess for postoperative time interval where NSAID medications may be safely administered without increasing incidence of postoperative bleeding events.

We propose a study comparing impact of maximally-dosed ibuprofen (10 mg/kg every 6 hours) versus maximally-dosed acetaminophen (15 mg/kg every 6 hours) on postoperative pain and bleeding when administered for four days (short-course) to children age 2-18 undergoing tonsillectomy with or without adenoidectomy. We believe that a four-day course of medication is appropriate given that the majority of post-tonsillectomy bleeding events occurred on day 6 and the half-life of ibuprofen is such that platelet function returns to baseline within 24 hours of drug discontinuation20. We hypothesize that children aged 2-18 receiving short-course ibuprofen following tonsillectomy will not have increased incidence of bleeding when compared to patients receiving acetaminophen postoperatively. A study definitively documenting safety and efficacy of short-course NSAID administration following tonsillectomy in children would affect our own standard of care as well as overall clinical practice guidelines surrounding this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ages 2-18 undergoing tonsillectomy with or without adenoidectomy by electrocautery alone for all indications
* Patients with complex medical conditions and craniofacial abnormalities will be included.
* Family must understand and be able to read English.
* Only patients who are not pregnant will be included.
* Informed consent and, child assent (when appropriate) will be required for enrollment. Patients will provide signed and dated informed consent form.
* Subjects will be willing and able to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* Patients with a known personal or family history of a bleeding disorder.
* Patients with a history of asthma, kidney or liver problems.
* Patients with tonsillectomy or adenoidectomy performed using a cold knife technique, microdebrider, coblation or plasma knife.
* Patients on NSAIDs for other medical conditions or those who have taken NSAIDs within 1 week of surgery
* Patients with allergy to aspirin or other NSAIDs, acetaminophen, Red Dye #40 or Red Dye #33
* Patients found to be pregnant will be excluded from participation. Pregnancy testing using urine beta-HCG will be performed on all children > 13 years of age, or those younger than 13 who are menstruating; this is the testing protocol used at the Children's Hospital of Boston.

Patients unwilling to enroll in the study will have the tonsillectomy with or without adenoidectomy performed according to current practice standards.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Post-tonsillectomy bleeding within 14 days of surgery. | Within 14 days of surgery
  This will be classified by timing (<24 hours vs. 24 hours or more) and severity (level 1: bleeding by history alone; level 2: objective bleeding requiring hospital admission and observation; level 3: objective bleeding requiring operative intervention). Bleeding events will be documented during postoperative visit at two weeks as well as through medical record review.

SECONDARY OUTCOMES:
Post-tonsillectomy pain control data through 14 days of surgery | Through 14 days of surgery
  Post-tonsillectomy pain control data through 14 days of surgery. Patients and family members will receive validated pain control questionnaires to be filled out every day for the first 14 days following surgery (see Appendix ).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Hartnick, MD, Principal Investigator — Massachusetts Eye and Ear
Locations (5):
- United States (5):
  - Rady's Children's Hospital, San Diego, California
  - Emory University and Children's Healthcare of Atlanta, Atlanta, Georgia
  - Case Western University- Raimbow Babies and Children's, Cleveland, Ohio
  - Portsmouth Naval Hospital, Portsmouth, Virginia
  - Madigan Army Hospital, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baugh RF, Archer SM, Mitchell RB, Rosenfeld RM, Amin R, Burns JJ, Darrow DH, Giordano T, Litman RS, Li KK, Mannix ME, Schwartz RH, Setzen G, Wald ER, Wall E, Sandberg G, Patel MM; American Academy of Otolaryngology-Head and Neck Surgery Foundation. Clinical practice guideline: tonsillectomy in children. Otolaryngol Head Neck Surg. 2011 Jan;144(1 Suppl):S1-30. doi: 10.1177/0194599810389949. PMID 21493257
- [Background] Boss EF, Marsteller JA, Simon AE. Outpatient tonsillectomy in children: demographic and geographic variation in the United States, 2006. J Pediatr. 2012 May;160(5):814-9. doi: 10.1016/j.jpeds.2011.11.041. Epub 2011 Dec 17. PMID 22183449
- [Background] Alexander NS, Schroeder JW Jr. Pediatric obstructive sleep apnea syndrome. Pediatr Clin North Am. 2013 Aug;60(4):827-40. doi: 10.1016/j.pcl.2013.04.009. PMID 23905822
- [Background] Schwengel DA, Dalesio NM, Stierer TL. Pediatric obstructive sleep apnea. Anesthesiol Clin. 2014 Mar;32(1):237-61. doi: 10.1016/j.anclin.2013.10.012. PMID 24491659
- [Background] Spicuzza L, Leonardi S, La Rosa M. Pediatric sleep apnea: early onset of the 'syndrome'? Sleep Med Rev. 2009 Apr;13(2):111-22. doi: 10.1016/j.smrv.2008.07.001. Epub 2008 Dec 5. PMID 19058983
- [Background] Randall DA, Hoffer ME. Complications of tonsillectomy and adenoidectomy. Otolaryngol Head Neck Surg. 1998 Jan;118(1):61-8. doi: 10.1016/S0194-5998(98)70376-6. PMID 9450830
- [Background] Subramanyam R, Varughese A, Willging JP, Sadhasivam S. Future of pediatric tonsillectomy and perioperative outcomes. Int J Pediatr Otorhinolaryngol. 2013 Feb;77(2):194-9. doi: 10.1016/j.ijporl.2012.10.016. Epub 2012 Nov 16. PMID 23159321
- [Background] Tan GX, Tunkel DE. Control of Pain After Tonsillectomy in Children: A Review. JAMA Otolaryngol Head Neck Surg. 2017 Sep 1;143(9):937-942. doi: 10.1001/jamaoto.2017.0845. PMID 28662233
- [Background] Cohen N, Sommer DD. Post-tonsillectomy pain control: consensus or controversy? Pain Manag. 2016;6(1):31-7. doi: 10.2217/pmt.15.58. Epub 2015 Dec 17. PMID 26678541
- [Background] Moir MS, Bair E, Shinnick P, Messner A. Acetaminophen versus acetaminophen with codeine after pediatric tonsillectomy. Laryngoscope. 2000 Nov;110(11):1824-7. doi: 10.1097/00005537-200011000-00011. PMID 11081593
- [Background] Isaacson G. Pediatric tonsillectomy: an evidence-based approach. Otolaryngol Clin North Am. 2014 Oct;47(5):673-90. doi: 10.1016/j.otc.2014.06.011. Epub 2014 Aug 7. PMID 25213277
- [Background] Isaacson G. Tonsillectomy care for the pediatrician. Pediatrics. 2012 Aug;130(2):324-34. doi: 10.1542/peds.2011-3857. Epub 2012 Jul 2. PMID 22753552
- [Background] Romsing J, Hertel S, Harder A, Rasmussen M. Examination of acetaminophen for outpatient management of postoperative pain in children. Paediatr Anaesth. 1998;8(3):235-9. doi: 10.1046/j.1460-9592.1998.00768.x. PMID 9608969
- [Background] Zubieta JK, Smith YR, Bueller JA, Xu Y, Kilbourn MR, Jewett DM, Meyer CR, Koeppe RA, Stohler CS. Regional mu opioid receptor regulation of sensory and affective dimensions of pain. Science. 2001 Jul 13;293(5528):311-5. doi: 10.1126/science.1060952. PMID 11452128
- [Background] Sadhasivam S, Myer CM 3rd. Preventing opioid-related deaths in children undergoing surgery. Pain Med. 2012 Jul;13(7):982-3; author reply 984. doi: 10.1111/j.1526-4637.2012.01419.x. Epub 2012 Jun 13. PMID 22694279
- [Background] Whittaker MR. Opioid use and the risk of respiratory depression and death in the pediatric population. J Pediatr Pharmacol Ther. 2013 Oct;18(4):269-76. doi: 10.5863/1551-6776-18.4.269. PMID 24719587
- [Background] Burian M, Geisslinger G. COX-dependent mechanisms involved in the antinociceptive action of NSAIDs at central and peripheral sites. Pharmacol Ther. 2005 Aug;107(2):139-54. doi: 10.1016/j.pharmthera.2005.02.004. Epub 2005 Apr 19. PMID 15993252
- [Background] Goldenberg NA, Jacobson L, Manco-Johnson MJ. Brief communication: duration of platelet dysfunction after a 7-day course of Ibuprofen. Ann Intern Med. 2005 Apr 5;142(7):506-9. doi: 10.7326/0003-4819-142-7-200504050-00009. PMID 15809462
- [Background] Rainsford KD. Ibuprofen: pharmacology, efficacy and safety. Inflammopharmacology. 2009 Dec;17(6):275-342. doi: 10.1007/s10787-009-0016-x. Epub 2009 Nov 21. PMID 19949916
- [Background] St Charles CS, Matt BH, Hamilton MM, Katz BP. A comparison of ibuprofen versus acetaminophen with codeine in the young tonsillectomy patient. Otolaryngol Head Neck Surg. 1997 Jul;117(1):76-82. doi: 10.1016/S0194-59989770211-0. PMID 9230328
- [Background] Kelly LE, Sommer DD, Ramakrishna J, Hoffbauer S, Arbab-Tafti S, Reid D, Maclean J, Koren G. Morphine or Ibuprofen for post-tonsillectomy analgesia: a randomized trial. Pediatrics. 2015 Feb;135(2):307-13. doi: 10.1542/peds.2014-1906. PMID 25624387
- [Background] Harley EH, Dattolo RA. Ibuprofen for tonsillectomy pain in children: efficacy and complications. Otolaryngol Head Neck Surg. 1998 Nov;119(5):492-6. doi: 10.1016/S0194-5998(98)70107-X. PMID 9807075
- [Background] Lewis SR, Nicholson A, Cardwell ME, Siviter G, Smith AF. Nonsteroidal anti-inflammatory drugs and perioperative bleeding in paediatric tonsillectomy. Cochrane Database Syst Rev. 2013 Jul 18;2013(7):CD003591. doi: 10.1002/14651858.CD003591.pub3. PMID 23881651